CLINICAL TRIAL: NCT01008644
Title: Do Plasma Osmolality Changes Influence Ventilation, and Are There Gender Differences?
Brief Title: Do Changes in Plasma Osmolality Influence Ventilation?
Acronym: OSM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vibeke Moen (Other)
Responsible Party: Sponsor-Investigator, Vibeke Moen, MD, Department of Anaesthesia, Kalmar County Hospital
Organization: Kalmar County Hospital (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: M-126-09
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Hyponatraemia; Hypernatraemia
Keywords: carbon dioxide; ventilation; gender; osmolality; menstruation cycle
MeSH Terms: conditions — Hyponatremia; Hypernatremia; Respiratory Aspiration; Coitus | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Experimental): The subjects will receive saline 3% intravenously for 2 hours, the volume calculated as 0.1 ml/kg/min.
  Interventions: Other: Water; Other: Saline 3%
- Water (Experimental): The subjects will drink tap water for 2 hours, the volume calculated as 20ml/kg/hour
  Interventions: Other: Water; Other: Saline 3%

INTERVENTIONS:
Other: Water — The subjects will drink tap water for 2 hours, volume calculated according to weight: 20ml/kg/hour.
  Other Names: saline 3%
Other: Saline 3% — The subjects will receive saline 3% intravenously for 2 hours, the volume calculated as 0.1 ml/kg/min

SUMMARY:
Primary hypothesis: osmolality changes influence the sensitivity of the respiratory center to carbon dioxide, hyponatraemia causing hyperventilation, and hypernatraemia depressing ventilation.

Secondary hypothesis: There are gender differences in the sensitivity to osmolality changes.

10 women and 10 men will on different occasions drink water or receive hypertonic saline intravenously, in order to lower or increase plasma osmolality. The women will participate during both faces of the menstruation cycle. On each occasion the subject´s sensitivity to carbon dioxide will be tested, and blood samples will be drawn for analysis of blood gases,electrolyte and osmolality.Subjects who interrupt participation before completion of all planned occasions, will be substituted, so that 10 subjects of either sex will have participated as planned. All results from all participants will be analyzed.

DETAILED DESCRIPTION:
Healthy volunteers will on different occasions be subject to reduced plasma osmolality caused by drinking water, and increased osmolality caused by intravenous infusion of hypertonic saline.Before and after each osmolality change, sensitivity to carbon dioxide will be tested by partial rebreathing through a so called Bain-system. Throughout the whole experiment heart rate, blood pressure and oxygen saturation will be recorded.Blood samples will be collected before each rebreathing test and every 20 minutes during the two hours of water or salt load. Urine will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Females with regular menstruations, males

Exclusion Criteria:

* Consumption of nicotine, BMI > 26,
* pregnancy,any hormone treatment,
* treatment with diuretics,
* diabetes or kidney disease,
* BMI > 26,

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
pCO2 | ten minutes
  pCO2,osmolality and sensitivity to CO2 will be recorded 10 minutes before before and 10 minutes after administering water or saline for two hours.The results will be analyzed for differences before and after osmolality changes in every single individual, and differences between females in luteal or follicular menstruation phase.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Irestedt. MD PhD, Study Director — Department of Anaesthesia and Intensive Care , Karolinska University Hospital, Stockholm
Locations (1):
- Department of Anaesthesia and Intensive care, Kalmar County Hospital, Kalmar, Kalmar County, Sweden

REFERENCES:
- [Background] Jennings DB. The physicochemistry of [H+] and respiratory control: roles of PCO2, strong ions, and their hormonal regulators. Can J Physiol Pharmacol. 1994 Dec;72(12):1499-512. doi: 10.1139/y94-216. PMID 7736341
- [Background] Weissgerber TL, Wolfe LA, Hopkins WG, Davies GA. Serial respiratory adaptations and an alternate hypothesis of respiratory control in human pregnancy. Respir Physiol Neurobiol. 2006 Aug;153(1):39-53. doi: 10.1016/j.resp.2005.09.004. Epub 2005 Nov 28. PMID 16311079
- [Background] Heenan AP, Wolfe LA. Plasma osmolality and the strong ion difference predict respiratory adaptations in pregnant and nonpregnant women. Can J Physiol Pharmacol. 2003 Sep;81(9):839-47. doi: 10.1139/y03-072. PMID 14614519